CLINICAL TRIAL: NCT02940041
Title: Concordance Between Gynaecologic Sonography Amd Pelvic MRI for the Pre-surgical Diagnosis of Uterine Mesenchymal Malignant Tumors
Brief Title: Concordance Between Sonography Amd MRI for Presurgical Diagnosis of Uterine Mesenchymal Malignant Tumors
Acronym: CERTUM
Status: Terminated | Type: Observational
Why Stopped: Not enough patients included
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-TUM-2016-30
Record Dates: First submitted 2016-10-18; First posted 2016-10-20 (Estimated); Last update posted 2023-12-26 (Actual); Status verified 2023-11

CONDITIONS: Leiomyoma; Leiomyosarcoma
Keywords: Diagnosis; Sonography; Magnetic Resonance
MeSH Terms: conditions — Leiomyoma; Leiomyosarcoma; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Pre-surgical diagnosis of uterine malignant tumors — All patientes who fit inclusion criteria will undergo a gynecologic sonography, pelvic MRI, determination of LDH, as in regular practice. No additional interventions will be done to any patient.

SUMMARY:
Determine the concordance between gynaecological sonography and pelvic MRI for the pre-surgical diagnosis of uterine malignant tumors.

DETAILED DESCRIPTION:
The hypothesis that will be evaluated with this study is the concordance between the sonographic assessment following the terms and definitions to describe uterine pathology proposed by Morphological Uterus Sonographic Assessment (MUSA) and the pelvic MRI for the pre-surgical diagnosis of malignant mesenchymal uterine tumors in patients affected of symptomatic leiomyomas with clinical or sonographic risk factors for atypical fibroids.

If both explorations have the same efficiency for the diagnosis, one of those should be avoided, diminishing the costs and surgery delay for these patients.

Those women with uterine leiomyoma who present >2 risk factors for uterine malignant mesenchymal tumors OR with sonographic criteria for atypical leiomyoma will be invited to participate in the study and will sign the informed consent.

After this first visit, the patient will undergo a gynecological sonography, serum lactate dehydrogenase (LDH) determination and a pelvic MRI, as it is done in our regular clinical practice.

All explorations will be performed in the same study center and will be done by independent physicians.

Then patients included will be addressed to a second visit to explain the results and surgery planning if it's needed.

One month after the surgery, one last visit will be conducted to perform a post-surgery control and give the final anatomo-pathological report of the surgery specimen. All data will be entered in the database for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Accept to participate in the study
* uterine leiomyomas who have >2 risk factors for mesenchymal uterine malignant tumor OR sonographic suspicion of atypical leiomyoma.

Exclusion Criteria:

* < 18 years
* Not being capable of understanding the study design

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women over 18 years old with uterine leiomyomas who have >2 risk factors for mesenquimal uterine malignant tumor OR sonographic suspicion of atypical leiomyoma.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Concordance Between Gynaecologic Sonography Amd Pelvic MRI | We expect to recruit 50 patients in 1 year period

SECONDARY OUTCOMES:
Determine sensibility for sonographic and MRI specific parameters on diagnosis uterine malignant tumors | We expect to recruit 50 patients in 1 year period
  Sonographic parameters : Undefined margins, Unique or multiple lesions, Size and Color-score (1,2,3,4) MRI parameters: Heterogenic or intermediate T2 Signal intensity , High or Intermediate b1000 signal, Apparent diffusion parameter <1.23, heterogeneous contrast catchment

IPD SHARING:
Plan to Share IPD: Yes